CLINICAL TRIAL: NCT02638584
Title: Effects of Ilaprazole 20mg on Ulcer Healing Rate and Prevention of Gastrointestinal Bleeding in the Patients Undergone Endoscopic Submucosal Dissection(ESD) for Gastric Adenoma or Early Gastric Cancer.
Brief Title: Effects of Ilaprazole on Ulcer Healing Rate and Prevention of Gastrointestinal Bleeding in the Patients Undergone ESD.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUMC-ILA01
Record Dates: First submitted 2015-12-14; First posted 2015-12-23 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2018-08

CONDITIONS: Gastric Cancer
Keywords: Ilaprazole; Gastric Adenoma; Early Gastric Cancer; Endoscopic Submucosal Dissection
MeSH Terms: conditions — Stomach Neoplasms | interventions — ilaprazole; Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ilaprazole (Experimental): Ilaprazole tab 10mg, 2 tablets once daily for 8 weeks.
  Interventions: Drug: Ilaprazole
- Rabeprazole (Active Comparator): Rabeprazole tab 20mg, 1 tablet once daily for 8 weeks.
  Interventions: Drug: Rabeprazole

INTERVENTIONS:
Drug: Ilaprazole — Ilaprazole 10mg 2tablets once a day(1 times / day), before breakfast
  Other Names: Ilaprazole(Noltec®)
  Arms: Ilaprazole
Drug: Rabeprazole — Rabeprazole 20mg 1tablets once a day(1 times / day), before breakfast
  Other Names: Pariet®
  Arms: Rabeprazole

SUMMARY:
This study compared Ulcer healing rate of Ilaprazole 20mg or Rabeprazole 20mg in the patients undergone Endoscopic Submucosal Dissection for Gastric Adenoma or Early Gastric Cancer and investigated Prevention of gastrointestinal bleeding.

DETAILED DESCRIPTION:
This study is a Multicenter, Randomized, Parallel and Prospective study to compare Ulcer healing rate of Ilaprazole 20mg or Rabeprazole 20mg in the patients undergone Endoscopic Submucosal Dissection for Gastric Adenoma or Early Gastric Cancer and to investigate Prevention of gastrointestinal bleeding.

Participants are defined as persons who underwent a Endoscopic Submucosal Dissection for Gastric Adenoma or Early Gastric Cancer. For 8 weeks, Participants treated as Ilaprazole 20mg or Rabeprazole 20mg once a day. After treatment, The ulcer healing rate was evaluated by Endoscopy at 4, 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 19 year old ≤ Male or female < 85 year old
* Subject who underwent Endoscopic Submucosal Dissection for Gastric Adenoma or Early Gastric Cancer
* Subject who agrees to participate and spontaneously sign the Informed consent form(ICF).

Exclusion Criteria:

* Known hypersensitivity to any component of ilaprazole
* Subjects who are taking contraindicated medications(ex. atazanavir) for experimental and concomitant drug.
* Subjects with abnormal levels in the laboratory tests

  * Total Bilirubin, Creatinine> 1.5 times upper limit of normal
  * Alanine transaminase(ALT), Aspartate transaminase(AST), Alkaline phosphatase, Blood urea nitrogen(BUN)> 2 times upper limit of normal
* Subjects diagnosed with other cancer within 5 years other than stomach cancer.
* Subjects with a history of Zollinger-Ellison syndrome, Barrett's esophagus, primary esophageal motility abnormality, esophageal strictures, pancreatitis, malabsorption, severe cardiovascular or pulmonary disease
* Subjects with a history of major surgery that can affect gastric acid secretion.
* Subjects should continue taking the following medicine during the study period : anticholinergics, promoting motility agents, prostaglandin analogs, sucralfate, aspirin, steroid, NSAIDs drug
* Subjects with uncontrolled organ failure (liver dysfunction, renal dysfunction)
* Pregnant and/or lactating women
* Subjects participating in a clinical trial before another trial within 30 days
* Inconsistency judged subject by researcher

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2015-12; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
The Ulcer healing rate after endoscopic submucosal dissection | participants will be followed at 8 weeks

SECONDARY OUTCOMES:
The rate of Ulcer size reduction as assessed by measurements of ulcer size change. | at 8 weeks after treatment
  The rate of Ulcer size reduction(Δ) : [(Initial ulcer size) - (Ulcer size at 8 weeks)] / (Initial ulcer size)
The quality of ulcer healing as evaluated by the observation of investigator at tracking endoscopy. | at 8 weeks after treatment
  Apply 0.15% Indigo carmine to scarring of the ulcer and Describe the pattern of the scar as flat, nodular or intermediate at tracking endoscopy.
The evaluation of symptom score as assessed by the Korean Gastrointestinal Symptom Rating Scale questionnaire. | at 8 weeks after treatment
  The Korean Gastrointestinal Symptom Rating Scale questionnaire measured the patient's symptom degree.

CONTACTS AND LOCATIONS:
Overall Officials: ChangSeok Bang, MD, PhD, Principal Investigator — HALLYM UNIVERSITY MEDICAL CENTER, Chuncheon Sacred Heart Hospital
Locations (1):
- HALLYM UNIVERSITY MEDICAL CENTER, Chuncheon Sacred Heart Hospital, Chuncheon, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
not yet decided

REFERENCES:
- [Derived] Bang CS, Shin WG, Seo SI, Choi MH, Jang HJ, Park SW, Kae SH, Yang YJ, Shin SP, Baik GH, Kim HY. Effect of ilaprazole on the healing of endoscopic submucosal dissection-induced gastric ulcer: randomized-controlled, multicenter study. Surg Endosc. 2019 May;33(5):1376-1385. doi: 10.1007/s00464-018-6412-9. Epub 2018 Aug 30. PMID 30167954